CLINICAL TRIAL: NCT02750423
Title: Neurologic Injury AAR: Neurologic Injury Following Aortic Arch Replacement: A Comparison of Two Different Cerebral Protection Strategies (A Pilot Study)
Brief Title: Neurologic Injury Following Aortic Arch Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Bradley Leshnower, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087270
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Aortic Arch Replacement; Hemi Arch Replacement
Keywords: Cardiology; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHCA+RCP (Active Comparator): Participants undergoing ascending aortic and hemiarch replacement will receive deep hypothermic circulatory arrest and retrograde cerebral perfusion (DHCA+RCP).
  Interventions: Procedure: DHCA+RCP
- MHCA+uSACP (Active Comparator): Participants undergoing ascending aortic and hemiarch replacement will receive moderate hypothermic circulatory arrest and unilateral selective antegrade cerebral perfusion (MHCA+uSACP).
  Interventions: Procedure: MHCA + SACP

INTERVENTIONS:
Procedure: DHCA+RCP — During deep hypothermic circulatory arrest and retrograde cerebral perfusion (DHCA+RCP) the participant is placed on cardiopulmonary bypass (heart-lung machine) and their body temperature is lowered to a range of 14-18 °C. Once the goal temperature has been achieved, the circulation is stopped and aortic arch replacement is performed in a bloodless surgical field. Blood will be pushed to the brain through arterial vessels, much like the natural blood flow pattern. Once the aortic arch repair is complete, cardiopulmonary bypass is reinstituted, the participant is rewarmed, and separated from cardiopulmonary bypass.
  Arms: DHCA+RCP
Procedure: MHCA + SACP — During moderate hypothermic circulatory arrest and unilateral selective antegrade cerebral perfusion (MHCA + SACP) the participant is placed on cardiopulmonary bypass (heart-lung machine0 and the native blood flow to the brain is temporarily suspended. The body is cooled to temperatures of ≤28°C and blood is administered to the brain via an artery in the neck during the period of arch reconstruction. Once the aortic arch repair is complete, cardiopulmonary bypass is reinstituted, the participant is rewarmed, and separated from cardiopulmonary bypass.
  Arms: MHCA+uSACP

SUMMARY:
Investigators are seeking to learn how well different cooling temperatures along with different blood flow pathways to the brain reduce the risk of injury to the brain in participants planning to undergo elective aortic arch and hemiarch surgery. Participants will be randomized to receive a cerebral protection strategy of either: deep hypothermic circulatory arrest and retrograde cerebral perfusion (DHCA+RCP) or moderate hypothermic circulatory arrest and unilateral selective antegrade cerebral perfusion (MHCA+uSACP). Evidence of neurologic injury will be assessed with neurologic exams, neurocognitive tests, MRI imaging of the brain and measurement of plasma S-100 levels during post operative follow ups.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the impact of the two most commonly employed methods of cerebral protection upon mitigating neurologic injury in participants planning to undergo elective aortic arch and hemiarch surgery. Participants will be recruited from patients undergoing ascending aortic and hemiarch replacement using hypothermic circulatory arrest at Emory University Hospital and Emory Saint Joseph's Hospital. Participants will be randomized to receive a cerebral protection strategy of either: deep hypothermic circulatory arrest and retrograde cerebral perfusion (DHCA+RCP) or moderate hypothermic circulatory arrest and unilateral selective antegrade cerebral perfusion (MHCA+uSACP). Evidence of neurologic injury will be assessed with neurologic exams, neurocognitive tests, MRI imaging of the brain and measurement of plasma S-100 levels during post operative follow up. Follow up visits will be conducted at Days 1, 3, 7, and 180 post operation.

ELIGIBILITY:
Inclusion Criteria:

Patients at Emory University Hospital and Emory Saint Joseph's Hospital planning to undergo:

* Elective surgical replacement of the ascending aorta and proximal ("hemiarch") using hypothermic circulatory arrest
* Concomitant cardiac procedures (e.g valve replacement, coronary artery bypass, etc.) in addition to ascending aortic and hemiarch replacement
* Any of the following cannulation and cerebral protection strategies:

  1. Right axillary artery cannulation, deep hypothermic circulatory arrest, retrograde cerebral perfusion
  2. Right axillary artery cannulation, moderate hypothermic circulatory arrest, unilateral selective antegrade cerebral perfusion

Exclusion Criteria:

* Undergoing total arch replacement
* Undergoing hemiarch replacement without the use of hypothermic circulatory arrest
* Undergoing hemiarch replacement using hypothermic circulatory arrest with a method of cerebral protection not listed in the Eligibility Criteria.
* Pregnant women or women who are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Stroke | Duration of Study (Up to 180 days)
  The number of participants with a new focal neurologic deficit lasting greater than 24 hours that is confirmed by radiographic evidence of infarction.
Incidence of Transient Ischemic Attack (TIA) | Duration of Study (Up to 180 days)
  The number of participants with a new focal neurologic symptom lasting less than 24 hours without radiographic evidence of infarction.
Rate of Neurologic Injury assessed by Magnetic Resonance Imaging (MRI) | Duration of Study (Up to 180 days)
  The number of participants with evidence of neurologic injury assessed by MRI.
Change in Verbal Memory Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The verbal memory test measures how many words participants can keep in short term memory at once. A higher score indicates better short term memory.
Change in Visual Memory Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The visual memory test measures how many items a participant can keep in short term memory at once. A higher score indicates better short term memory.
Change in Finger Tapping Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The finger-tapping test (FTT) is a neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination. During administration, the participant's palm should be immobile and flat on the board, with fingers extended, and the index finder placed on the counting device. One hand at a time, participants tap their index finger on the lever as quickly as possible within a 10-s time interval, in order to increase the number on the counting device with each tap.
Change in Symbol Digit Coding Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The Digit symbol substitution test (DSST) is a neuropsychological test sensitive to brain damage, dementia, age and depression. It consists of nine digit-symbol pairs followed by a list of digits.Under each digit the participant should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured.
Change in Stroop Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The Stroop effect is a demonstration of interference in the reaction time of a task. Participants will be asked the name of a color printed in a color not denoted by the name. Naming the color of the word takes longer and is more prone to errors than when the color of the ink matches the name of the color.
Change in Shifting Attention Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The Shifting Attention Test measures a participant's executive functions (rules, categories, rapid decision making) or their ability to shift from one instruction set to another quickly and accurately.
Change in Continuous Performance Test Score | Post Operative Visit Day 1, Post Operative Visit Day 180
  The continuous performance test measures a participant's sustained and selective attention. Sustained attention is the ability to maintain a consistent focus on some continuous activity or stimuli, and is associated with impulsivity. Selective attention is the ability to focus on relevant stimuli and ignore competing stimuli. This skill is associated with distractibility.[1]

SECONDARY OUTCOMES:
Incidence of Temporary Neurologic Deficit (TND) | Duration of Study (Up to 180 days)
  The number of participants with a reversible, non-focal clinical neurologic injury without radiographic evidence of infarction.
Change in Serum S-100 Levels | Post Operative Visit Day 1, Post Operative Visit Day 180
  Serum S-100 is a biomarker for neurologic injury found in blood serum.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Leshnower, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia